CLINICAL TRIAL: NCT00331253
Title: A 54-WEEK, PHASE 2, MULTICENTER, MASKED, RANDOMIZED, CONTROLLED TRIAL TO ESTABLISH THE SAFETY AND EFFICACY OF INDOCYANINE GREEN-MEDIATED PHOTOTHROMBOSIS (i-MP) FOR THE TREATMENT OF PATIENTS WITH NEOVASCULAR AGE-RELATED MACULAR DEGENERATION.
Brief Title: Treatment of Patients With Neovascular AMD Using Indocyanine Green-Mediated Photothrombosis (i-MP).
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Opto Eletronica S.A. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 001/04/i-MP
Record Dates: First submitted 2006-05-26; First posted 2006-05-29 (Estimated); Last update posted 2007-04-27 (Estimated); Status verified 2007-04

CONDITIONS: Maculopathy, Age-Related
Keywords: Indocyanine Green-Mediated Photothrombosis; Neovascular; Age-Related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Indocyanine Green-Mediated Photothrombosis

SUMMARY:
To establish the safety and efficacy of indocyanine green-mediated photothrombosis (i-MP) for the treatment of patients with neovascular age-related macular degeneration.

DETAILED DESCRIPTION:
Comparative, controlled, multicenter, masked, randomized study, three parallel groups, comparing the Indocyanine Green-Mediated Photothrombosis to two control groups, for the treatment of neovascular Age-Related Macular Degeneration.

Only patients matching the following criteria are eligible:

A. BCVA worse than 20/80 and neovascular complex with some component of occult CNV as defined by the fluorescein angiography, or; B. BCVA worse than 20/80 and neovascular complex with total area of CNV (classic and occult) by fluorescein angiography occupying an area lesser than 50% of the neovascular complex, or; C. BCVA worse than 20/200 and neovascular complex with some CNV (classic OR occult) by fluorescein angiography.

The eligibility of the patients will be assessed by an independent Centre of Interpretation after masked analysis.

Eligible patients will be allocated into one of the three study groups, randomized at 2:1:1 proportion:

Group 1: Treatment Procedure #1 = i-MP (ICG + Laser), at proportion of 2. In this group the patients will be submitted to endovenous infusion of ICG followed by irradiation with diode laser.

Group 2: Treatment Procedure #2 (Distilled water + Laser), at proportion of 1. In this group the patients will receive endovenous placebo infusion (distilled water) followed by irradiation with diode laser with same power utilized in Group 1.

Group 3: Treatment Procedure #3 (Distilled water + Sham Laser), at proportion of 1. In this group the patients will receive endovenous placebo infusion (distilled water) followed by simulated application of laser.

ELIGIBILITY:
Inclusion Criteria:

* Age over 50 years;
* Presence of at least 1 soft drusen in the macular region, associated or not to pigment alterations (hyper- or hypo-pigmentation), thus characterising AMD;
* Reduction of vision due exclusively to macular exudative processes resulting from the formation of associated choroidal neovascularisation (neovascular AMD);
* Patients presenting:
* Neovascular complexes characterised by presence of some occult CNV component in their formation by fluorescein angiography and BCVA worse than 20/80, OR;
* Neovascular complexes with total CNV (classic and occult) area by fluorescein angiography occupying an area lesser than 50% of the neovascular complex and BCVA worse than 20/80, OR;
* BCVA lesser than 20/200, regardless of the type of composition of the neovascular complex;
* Direct involvement of the avascular foveal zone by the neovascular complex;
* Informed Consent Form in writing and appropriately signed.

Exclusion Criteria:

* BCVA lesser than 20/400;
* Greatest linear dimension of the neovascular complex greater than 6000 (six thousand) micron;
* Previous Photodynamic Therapy (PDT);
* Thermal laser for the treatment of any CNV;
* Intra vitreous injection of corticosteroids or anti-angiogenic drugs;
* Opacities of the media that can significantly interfere on the VA, clinical ophthalmic assessment, documentation of the eye fundus and performance of laser therapy;
* Other causes of CNV such as pathologic myopia (spherical equivalent greater than 6 [six] spherical diopters and/or axial length greater than 26mm), angioid streaks, active uveitis, ocular presumed histoplasmosis and traumatic choroidal rupture;
* CNV associated to serous/sero hemorrhagic RPED (vascular RPED / hemorrhagic RPED);
* Absence of identifiable CNV by fluorescein angiography (massive presence of thick blood);
* CNV with absence of ICG uptake by ICG angiography despite the eligibility of the patient by clinical criteria and fluorescein angiography;
* Intraocular surgery undertaken in the last 3 months;
* Posterior vitrectomy or retinopexy with scleral introflexion, at any time;
* Severe form of non-proliferative Diabetic Retinopathy;
* Acute ocular infection;
* Ionizing radiation treatment on the face, skull and neck region;
* Allergy to fluorescein or indocyanine green;
* Excessive known use of alcohol or drugs;
* Medical or psychological conditions which may impede the patient of completing the study or sing the Informed Consent Form;
* Significant uncontrolled disease which, in the opinion of the investigator, may exclude the patient from the study;
* Impediment or limited legal capability;
* Participation in other clinical study in the last 30 days. NOTE: Patients who have participated of any clinical study in the last 12 months, even though they had finished their participation prior to the last 30 days, will only be eligible to inclusion if the participation in the present protocol will bring clear benefit to the patient.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280
Dates: Start 2007-04; Study Completion 2008-12 (Estimated)

PRIMARY OUTCOMES:
Compare the groups in respect to proportion of eyes that lost less than 15 letters in ETDRS BCVA from baseline at week-54
Compare the groups in respect to proportion of eyes that did not present any loss in ETDRS BCVA (2 letters change) from baseline at week-54

SECONDARY OUTCOMES:
Compare the groups in respect to mean change in ETDRS BCVA
Compare the groups in respect to neovascular complex activity (size and CNV leaking area)

CONTACTS AND LOCATIONS:
Overall Officials: Elizeu Ramos, M.S., Study Director — Opto Eletrônica S.A.; Avila Marcos, MD, Principal Investigator — Universidade Federal de Goias
Locations (1):
- Universidade Federal de Goias, Goiânia, Goias/Go, Brazil